CLINICAL TRIAL: NCT00074178
Title: Combination Chemotherapy (Methotrexate, Cyclophosphamide, And Etoposide Phosphate) Delivered In Conjunction With Osmotic Blood-Brain Barrier Disruption (BBBD), With Intraventricular Cytarabine +/- Intra-Ocular Chemotherapy, In Patients With Primary Central Nervous System Lymphoma
Brief Title: Methotrexate, Cyclophosphamide, and Etoposide Phosphate Given With Osmotic Blood-Brain Barrier Disruption Plus Dexamethasone and Cytarabine in Treating Patients With Primary CNS Lymphoma
Acronym: Protocol-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000935; 5729-2 (Other: OHSU IRB (discontinued number)); ONC-99055-L (Other: OHSU Knight Cancer Institute); 935 (Other: OHSU eIRB); OHSU-5729-2 (Other: OHSU IRB (legacy number))
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Lymphoma
Keywords: primary central nervous system lymphoma; intraocular lymphoma
MeSH Terms: conditions — Lymphoma; Intraocular Lymphoma | interventions — Filgrastim; pegfilgrastim; Cyclophosphamide; Cytarabine; Dexamethasone; etoposide phosphate; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide phosphate
Drug: methotrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, cyclophosphamide, etoposide phosphate, dexamethasone, and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Osmotic blood-brain barrier disruption uses certain drugs to open the blood vessels around the brain and allow anticancer substances to be delivered directly to the brain. Giving methotrexate, cyclophosphamide, and etoposide phosphate with osmotic blood-brain barrier disruption plus dexamethasone and cytarabine may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of giving methotrexate, cyclophosphamide, and etoposide phosphate with osmotic blood-brain barrier disruption plus dexamethasone and cytarabine in treating patients who have primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity and efficacy of methotrexate, cyclophosphamide, and etoposide phosphate administered in conjunction with osmotic blood-brain barrier disruption and dexamethasone and cytarabine in patients with primary CNS lymphoma.

Secondary

* Determine the ability to recruit an adequate number of patients for this study.
* Compare progression-free and dementia-free survival with standard measures of overall survival, progression-free survival, disease-free survival, complete response rate, cognitive function, and quality of life of patients treated with this regimen.
* Determine the feasibility of conducting a future phase III study of this treatment regimen in this patient population.
* Correlate neuropsychological outcomes with neuroimaging (MRI) outcomes in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive methotrexate (MTX) intra-arterially over 10 minutes, cyclophosphamide IV over 10 minutes, and etoposide phosphate IV over 10 minutes on days 1 and 2 in conjunction with osmotic blood-brain barrier disruption. Patients also receive oral dexamethasone every 6 hours on days 2-15 (followed by a taper) and intraventricular or intrathecal cytarabine on day 14. Beginning 48 hours after the last dose of MTX, patients receive filgrastim (G-CSF)* subcutaneously once daily for 7-10 days or until blood counts recover. Treatment repeats every 4 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Alternatively, patients may receive a single dose of pegfilgrastim, administered 24 hours after the completion of chemotherapy

Patients with intraocular lymphoma also receive MTX intravitreally twice weekly until the vitreous is clear of cells by slit lamp exam and then weekly for 1 month and monthly for 1 year.

Quality of life is assessed at baseline, at 6 months, at the completion of treatment, and then every 6 months for 2 years and annually thereafter.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed intermediate- or high-grade primary CNS lymphoma by brain biopsy or cerebrospinal fluid or vitrectomy analysis
* No more than 90 days since diagnosis
* No systemic lymphoma NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 16 to 75

Performance status

* ECOG 0-3 OR
* Karnofsky 40-100%

Life expectancy

* Not specified

Hematopoietic

* Hematocrit at least 25% (transfusion allowed)
* WBC at least 2,500/mm^3
* Absolute granulocyte count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3 OR at least lower limit of normal (transfusion independent)

Hepatic

* Bilirubin no greater than 2.0 times upper limit of normal

Renal

* Creatinine clearance at least 30 mL/min

Cardiovascular

* Adequate cardiac function to tolerate general anesthesia

Pulmonary

* Adequate pulmonary function to tolerate general anesthesia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 2 months before and during study participation
* No other uncontrolled clinically significant confounding medical condition within the past 30 days
* No known allergy to study agents
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

  * Single-agent methotrexate administered within the past 14 days allowed

Endocrine therapy

* Not specified

Radiotherapy

* No prior cranial or spinal radiotherapy

Surgery

* Prior surgery or biopsy allowed

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Survival as measured by clinical and radiographic response at 5 years after study treatment

SECONDARY OUTCOMES:
Overall survival as measured by clinical and radiographic response
Progression-free survival as measured by clinical and radiographic response until tumor progression
Quality of Life (QOL) as measured by EORTC QOL before and after study treatment, every 6 months for 2 years, and then annually

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Neuwelt, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Oregon Health & Science University Cancer Institute, Portland, Oregon, United States